CLINICAL TRIAL: NCT04135417
Title: A Phase 2 Assessment of Humacyte's Human Acellular Vessel in Patients Needing Vascular Access for Dialysis
Brief Title: Safety and Efficacy Assessment of HAV in Patients Needing Vascular Access for Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PRO-V011
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Renal Failure; End Stage Renal Disease; Vascular Access; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HAV (Experimental): The HAV is a tissue-engineered vascular conduit (6mm diameter) for hemodialysis access in patients with end-stage renal disease. HAV for this study will be manufactured using the commercial manufacturing system.It will be implanted in the forearm or upper arm using standard vascular surgical techniques. All subjects will be required to start taking daily aspirin (75 or 325 mg) on Day 1 after surgical implantation of HAV unless they are already taking another antiplatelet agent. If low molecular weight heparin (LMWH) is administered post-operatively, aspirin or other antiplatelet agents should be initiated after stopping LMWH. Subjects who are known to be aspirin-sensitive should take another antiplatelet agent at the discretion of the Principal Investigator.
  Interventions: Biological: HAV

INTERVENTIONS:
Biological: HAV — Surgical implantation of the HAV and subsequent use of the implanted vascular conduit for hemodialysis vascular access.

SUMMARY:
This is a Phase 2, prospective, multicenter, open-label, single-arm study of the Human Acellular Vessel (HAV).

DETAILED DESCRIPTION:
This is a Phase 2, prospective, multicenter, open-label, single-arm study. Subjects who sign informed consent would undergo study-specific screening assessments within 45 days from the day of informed consent.

Eligible study subjects will receive a HAV and will be followed to 12 months post-implantation at routine study visits regardless of patency status. After 12 months, subjects with a patent HAV will be followed (while the HAV remains patent) for up to 2 years (24 months) post implantation at study visits every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with ESRD who are not, or who are no longer candidates for creation of an autologous AV fistula and therefore need placement of an AV graft in the arm (upper or forearm) for hemodialysis therapy.
2. Already established on hemodialysis
3. At least 18 years of age at Screening.
4. Suitable arterial and venous anatomy for implantation of straight or looped conduits in either the forearm or upper arm (not crossing the elbow).
5. Hemoglobin ≥ 8 g/dL and platelet count ≥ 100,000 cells/mm3 prior to Day 0 (within 45 days).
6. Other hematological and biochemical parameters within a range consistent with ESRD prior to Day 0 (within 45 days).
7. Normal clotting (international normalized ration [INR] ≤ 1.5 or prothrombin time ≤ 18 sec unless the patient is taking an anticoagulant for an approved indication at the time of HAV implantation.
8. Female subjects must be either:

   1. Of non-childbearing potential, which is defined as post-menopausal (at least 1 year without menses prior to Screening) or documented surgically sterile or post hysterectomy (at least 1 month prior to Screening)
   2. Or, of childbearing potential, in which case:

   i. Must have a negative serum or urine pregnancy test at Screening, and ii. Must agree to use at least one form of the following birth control methods for the duration of the study:

1. Established use of oral, injectable or implanted hormonal methods of contraception 2. Placement of an intrauterine device or intrauterine system 3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository 9. Subject, or legal representative, able to communicate effectively with investigative staff, competent and willing to give written informed consent, and able to comply with entire study procedures including all scheduled follow-up visits.

10. Life expectancy of at least 1 year.

Exclusion Criteria:

1. History or evidence of severe peripheral vascular disease in the intended arm for implantation.
2. Known or suspected central vein stenosis or conduit occlusion on the ipsilateral side of the planned implantation, unless the stenosis is corrected prior to HAV implantation.
3. Treatment with any investigational drug or device within 60 days prior to study entry (Day 0) or ongoing participation in a clinical trial of an investigational product.
4. Cancer that is actively being treated with a cytotoxic agent.
5. Documented hyper-coagulable state as defined as either:

   1. a biochemical diagnosis (e.g. Factor V Leiden, Protein C deficiency, etc.) - OR -
   2. a clinical history of thrombophilia as diagnosed by 2 or more spontaneous intravascular thrombotic events (e.g deep vein thrombosis, pulmonary embolism, etc.) within the 5 previous years.
6. Spontaneous or unexplained bleeding diathesis clinically documented within the last 5 years or a biochemical diagnosis (e.g. von Willebrand disease, etc.).
7. Active clinically significant immune-mediated disease, not controlled by maintenance immunosuppression.

   1. Low dose glucocorticoid therapy (e.g. up to 10 mg a day prednisone or prednisolone) is acceptable.
   2. High dose glucocorticoid therapy for treatment of autoimmune flare, or other inflammatory diseases is excluded.
   3. Patients using glucocorticoids for immunosuppression post-transplant to prevent against transplanted allograft rejection in the period post allograft failure are excluded.
   4. The following examples of immunosuppressive agents (or the like) are exclusionary for enrollment in this clinical trial:

   i. tacrolimus or FK506 [Prograf] ii. mycophenolate mofetil [Cellcept], iii. cyclosporine [Sandimmune or Gengraf] iv. Sirolimus administered systemically (Sirolimus in drug eluting stents is NOT an exclusion)
8. Anticipated renal transplant within 6 months.
9. Venous outflow from HAV cannot be placed more centrally than the venous outflow of any previous failed access on that extremity.
10. Active local or systemic infection (white blood cells [WBC] > 15,000 cells/mm3 at Screening). If the infection resolves, the subject must be at least 1 week post resolution of that infection before implantation.
11. Known serious allergy to planned antiplatelet agent.
12. Pregnant women, or women intending to become pregnant during the course of the trial.
13. Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the HAV.
14. Previous enrollment in this study or any other study with HAV.
15. Employees of Humacyte and employees or relatives of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamik Shamik, MD, Study Director — Humacyte, Inc.
Locations (2):
- Poland (2):
  - Szpital Kliniczny Przemienienia Pańskiego UM w Poznaniu, Klinika Chirurgii Ogólnej i Naczyń, Poznan
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Oddział Chirurgii Naczyniowej, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HAV (Continued in Description): The HAV is a tissue-engineered vascular conduit (6mm diameter) for hemodialysis access in patients with end-stage renal disease. HAV for this study will be manufactured using the commercial manufacturing system.It will be implanted in the forearm or upper arm using standard vascular surgical techniques. All subjects will be required to start taking daily aspirin (75 or 325 mg) on Day 1 after surgical implantation of HAV unless they are already taking another antiplatelet agent. If low molecular weight heparin (LMWH) is administered post-operatively, aspirin or other antiplatelet agents should be initiated after stopping LMWH. Subjects who are known to be aspirin-sensitive should take another antiplatelet agent at the discretion of the Principal Investigator.
  HAV: Surgical implantation of the HAV and subsequent use of the implanted vascular conduit for hemodialysis vascular access.
Period: Overall Study
Arm/Group | HAV (Continued in Description)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HAV (Continued in Description)
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.5 [38 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Poland | 30

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Subjects With Adverse Events Indicating Possible Mechanical Failure or Weakness of the HAV
Description: Frequency and severity of AEs of each patient will be documented
Time Frame: Up to 3 months post-implantation
Measure: Number; unit: participants
Arm/Group | HAV (Continued in Description)
Number analyzed (Participants) | 30
participants | 0

2. Primary Outcome: Number of Participants With Baseline Change of Panel Reactive Antibody (PRA) Value
Description: Assess changes in the PRA response (number of participants) over the 2 months after graft implantation
Time Frame: 2 months post implantation
Measure: Number; unit: participants
Arm/Group | HAV (Continued in Description)
Number analyzed (Participants) | 30
participants | 2

3. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI)
Description: Frequency and severity of all adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESI) of each patient will be documented.
Time Frame: Up to 3 months post-implantation
Measure: Number; unit: participants
Arm/Group | HAV (Continued in Description)
Number analyzed (Participants) | 30
participants
  All AEs | 12
  All SAEs | 7
  All AESI | 8

4. Primary Outcome: Number of Participants With Primary Patency, Primary Assisted Patency and Secondary Patency
Time Frame: 3 months post-implantation
Measure: Number; unit: participants
Arm/Group | HAV (Continued in Description)
Number analyzed (Participants) | 30
participants
  Loss of primary patency at Month 3 | 1
  Loss of primary assisted patency at Month 3 | 1
  Loss of secondary patency at Month 3 | 0

5. Secondary Outcome: Number of Participants With Baseline Change of Panel Reactive Antibody (PRA) Value
Description: Assess changes in the PRA response (number of subjects) over the 12 months after graft implantation
Time Frame: 12 months post-implantation
Population: In total, 4 subjects (13%) had an increase in PRA levels from Baseline that remained elevated through Month 12.
Measure: Number; unit: participants
Arm/Group | HAV (Continued in Description)
Number analyzed (Participants) | 30
participants | 4

6. Secondary Outcome: Number of Participants With All AEs/SAEs
Description: Frequency and severity of AEs/SAE of each patient will be documented
Time Frame: Up to 12 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | HAV (Continued in Description)
Number analyzed (Participants) | 30
Participants
  Number of Participants with All AEs | 25
  Number of Participants with All SAEs | 19

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | HAV (Continued in Description)
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 19/30
Other Adverse Events (participants affected / at risk) | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HAV (Continued in Description) (N=30)
Bradycardia, Cardiac failure (Cardiac disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Bacterial sepsis, Bronchitis, C diff infection, Corona virus infection, continued in description (Infections and infestations) | 8 — Diabetic foot infection, Hematoma infection, Localized infection, Vascular access site infection
Anatomic stenosis, Fall, Vascular access site hematoma, continued in description (Injury, poisoning and procedural complications) | 12 — Vascular access site pseudoaneurysm, Vascular access site thrombosis
Ischemic stroke (Nervous system disorders) | 1
Brachiocephalic vein stenosis (Vascular disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HAV (Continued in Description) (N=30)
Ventricular tachycardia (Cardiac disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Implant site erythema (General disorders) | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Vascular stenosis (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT04135417/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT04135417/SAP_001.pdf